CLINICAL TRIAL: NCT05109091
Title: A Randomized, Double-Blind, Placebo-Controlled Study of ATH434 in Multiple System Atrophy
Brief Title: Study of ATH434 in Participants with Multiple System Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alterity Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATH434-201
Record Dates: First submitted 2021-10-22; First posted 2021-11-05 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy; ATH434; Neurodegenerative disease; Shy-Drager Syndrome; Movement disorders; Autonomic dysfunction; Synucleinopathies; Atypical parkinsonism
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases; Shy-Drager Syndrome; Movement Disorders; Primary Dysautonomias; Synucleinopathies | interventions — 8-hydroxyquinazolin-4(3H)-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ATH434 Arm 1 (Experimental)
  Interventions: Drug: ATH434 dose level 1
- ATH434 Arm 2 (Experimental)
  Interventions: Drug: ATH434 dose level 2
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH434 dose level 1 — ATH434 taken BID
  Other Names: PBT434
  Arms: ATH434 Arm 1
Drug: ATH434 dose level 2 — ATH434 taken BID
  Other Names: PBT434
  Arms: ATH434 Arm 2
Drug: Placebo — Placebo taken BID
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of ATH434 in participants with Multiple System Atrophy

ELIGIBILITY:
Inclusion Criteria:

1. Participant has clinical features of parkinsonism.
2. Participant has evidence of orthostatic hypotension and/or bladder dysfunction.
3. Participant has ataxia and/or pyramidal signs on neurological examination.
4. Participant is ambulatory.
5. Participant has biomarker evidence of MSA in biologic fluid and on MRI.

Exclusion Criteria:

1. Participant has motor symptoms for > 4 years.
2. Participant has advanced disease, as indicated by frequent falls or choking.
3. Participant has structural brain abnormality on MRI.
4. Participant has any significant neurological disorder other than MSA.
5. Participant has an unstable medical or psychiatric illness.
6. Participant has a contraindication to, or is unable to tolerate, MRI or lumbar puncture.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Change in iron content as measured by brain MRI | Change from Baseline to Week 52

SECONDARY OUTCOMES:
Change in Neurofilament Light Chain Levels | Change from Baseline to Week 52
Change in Unified MSA Rating Scale (UMSARS) Score | Change from Baseline to Week 52
Change in SF-36 Score | Change from Baseline to Week 52

CONTACTS AND LOCATIONS:
Locations (23):
- United States (6):
  - University of California San Diego, La Jolla, California
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University Irving Medical Center, New York, New York
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (3):
  - St Vincent's Hospital (Sydney), Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- France (4):
  - CHU de Toulouse/Hôpital Pierre-Paul Riquet, Toulouse, Haute-Garonne
  - CHU de Bordeaux/Groupe Hospitalier Pellegrin, Bordeaux
  - CHU de Marseille/Hôpital de la Timone, Marseille
  - CHU/HU Pitié Salpêtrière, Paris, Île-de-France Region
- Italy (4):
  - IRCCS Istituto Delle Scienze Neurologiche di Bologna, Bologna, Bologna
  - Policlinico di Milano, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - AOU San Giovanni di Dio Ruggi d'Aragona, Salerno
- New Zealand (2):
  - New Zealand Brain Research Institute, Christchurch
  - Auckland City Hospital, Grafton
- United Kingdom (4):
  - University College London, London, England
  - Newcastle University, Newcastle upon Tyne, England
  - Salford Royal Hospital, Salford, England
  - Queen Elizabeth University Hospital, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No